CLINICAL TRIAL: NCT00701246
Title: Nutritional Anemia: Prevention and Treatment in Early Childhood
Brief Title: Treatment and Prevention of Anemia With Ferrous Sulfate Plus Folic Acid in Children in Goiania - Goias, Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Federal University of São Paulo (Other); Ministry of Health, Brazil (Other Government); Goiania Municipal Health Department (Unknown)
Responsible Party: Principal Investigator, Maria Claret Costa Monteiro Hadler, PhD., Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: FANUT 302004
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Anemia
Keywords: Anemia; Iron deficiency anemia; Infants; Children; Clinical trials; Ferrous sulfate; Folic acid; Daycare centers; Anaemia in children; born at term; non-twins; with parental approval for participation in the study; growth
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — ferrous sulfate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- I (Experimental): I Treatment: a daily dose (5 times a week) of either 4,2 mg/kg/day of ferrous sulfate + folic acid (50 mcg)
  Interventions: Drug: ferrous sulfate; Drug: folic acid
- II (Placebo Comparator): II Treatment of anemic children with 4,2 mg/kg/day of ferrous sulfate and folic acid placebo.
  Interventions: Drug: ferrous sulfate; Drug: placebo (folic acid)
- III (Experimental): Prevention of anemia in non-anemic children ( 5 times a week)- 1,4 mg/kg/day of ferrous sulfate and folic acid
  Interventions: Drug: ferrous sulfate; Drug: folic acid
- IV (Placebo Comparator): 1,4 mg/kg/day of ferrous sulfate plus folic acid placebo, five days a week.
  Interventions: Drug: ferrous sulfate; Drug: placebo (folic acid)

INTERVENTIONS:
Drug: ferrous sulfate
Drug: folic acid
  Arms: I; III
Drug: placebo (folic acid)
  Arms: II; IV

SUMMARY:
Iron deficiency anemia is the most common nutritional problem in the world.

The objectives of this study are:

* to evaluate the prevalence of anemia in children from 6 to 24 months of age and the therapeutic and prophylactic response to ferrous sulfate plus folic acid on hemoglobin levels.
* to compare the effect of folic acid supplementation with ferrous sulfate on the linear and weight growth of anemic and non-anemic

Study hypothesis:

* The ferrous sulfate plus folic acid can improve the response on hemoglobin levels.
* The folic acid supplementation with ferrous sulfate have effect on the linear and weight growth of anemic and non-anemic.

DETAILED DESCRIPTION:
Purpose

The objective of this study were:

* to assess the prevalence of anemia and the therapeutic and prophylactic response to ferrous sulfate and folic acid.
* to compare the effect of folic acid supplementation with ferrous sulfate on the linear and weight growth of anemic and non-anemic.

A double-blind, randomized, controlled clinical trial was conducted with 196 children 6 to 24 months of age enrolled in municipal daycare centers in Goiânia, Goias State, Brazil. The children were assigned to two treatment groups that received a daily dose (5 times a week) of either 4.2mg/kg/day of ferrous sulfate + folic acid (50μg) or 4.2mg/kg/day of ferrous sulfate + folic acid placebo. One of the prevention groups received 1.4mg/kg/day of ferrous sulfate + folic acid (50μg/day) and the other 1.4mg/kg/day of ferrous sulfate + folic acid placebo. Supplementation lasted approximately three months.

ELIGIBILITY:
Inclusion Criteria:

* from 6 to 24 months
* born at term
* non-twins
* with parental approval for participation in the study
* attending municipal daycare centers with mor than four children each

Exclusion Criteria:

* Children with special needs
* low birth weight (<2.500g)
* with growth-impairing heart diseases
* neurological syndromes
* sickle-cell anemia
* sickle-cell trait
* under treatment for anemia at the time of the first interview or screening performed by the pediatrician
* those no longer attending the daycare center
* the clinical trial excluded children with hemoglobin >=7 amd <=8g/dL.
* For the second objective: incomplete anthropometric surveys

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2005-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Iron status | Approximately three months

SECONDARY OUTCOMES:
Prevalence of anemia | Approximately three months

OTHER OUTCOMES:
Linear ad weight gain of anemic and non-anemic | Approximately three months
  Linear and weight gain of anemic and non-anemic observed by anthropometric surveys (Z-score for weight-for-age, Z-score for height-for-age, Z-score for weight-for-height, average monthly weight, monthly length gain, and gain of Z-scores for weight-for-age, height-for-age, weight-for-height)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Claret CM Hadler, PhD Sciences, Principal Investigator — Universidade Federal de Goias; Dirce M Sigulem, MD, PhD, Principal Investigator — Federal University of São Paulo; Maria de Fátima C Alves, PhD, Principal Investigator — Universidade Federal de Goias; Vinícius M Torres, MD, Principal Investigator — Vila São José Bento Cotolengo; Daniela AM Dias, MSc., Principal Investigator — Faculty of Nutrition of Federal University of Goias; Andréa Sugai, PhD., Principal Investigator — Faculty of Nutrition - Federal University of Goias
Locations (1):
- Universidade Federal de Goias, Goiânia, Goiás, Brazil

REFERENCES:
- [Background] Wieringa FT, Dijkhuizen MA, van der Ven-Jongekrijg J, West CE, Muhilal, van der Meer JW. Micronutrient deficiency and supplementation in Indonesian infants. Effects on immune function. Adv Exp Med Biol. 2003;531:369-77. doi: 10.1007/978-1-4615-0059-9_31. No abstract available. PMID 12916807
- [Background] Allen LH, Rosado JL, Casterline JE, Lopez P, Munoz E, Garcia OP, Martinez H. Lack of hemoglobin response to iron supplementation in anemic mexican preschoolers with multiple micronutrient deficiencies. Am J Clin Nutr. 2000 Jun;71(6):1485-94. doi: 10.1093/ajcn/71.6.1485. PMID 10837289
- [Background] Hadler MC, Juliano Y, Sigulem DM. [Anemia in infancy: etiology and prevalence]. J Pediatr (Rio J). 2002 Jul-Aug;78(4):321-6. Portuguese. PMID 14647764
- [Background] Hadler MC, Colugnati FA, Sigulem DM. Risks of anemia in infants according to dietary iron density and weight gain rate. Prev Med. 2004 Oct;39(4):713-21. doi: 10.1016/j.ypmed.2004.02.040. PMID 15351537
- [Background] Geltman PL, Meyers AF, Mehta SD, Brugnara C, Villon I, Wu YA, Bauchner H. Daily multivitamins with iron to prevent anemia in high-risk infants: a randomized clinical trial. Pediatrics. 2004 Jul;114(1):86-93. doi: 10.1542/peds.114.1.86. PMID 15231912
- [Background] Sazawal S, Black RE, Ramsan M, Chwaya HM, Stoltzfus RJ, Dutta A, Dhingra U, Kabole I, Deb S, Othman MK, Kabole FM. Effects of routine prophylactic supplementation with iron and folic acid on admission to hospital and mortality in preschool children in a high malaria transmission setting: community-based, randomised, placebo-controlled trial. Lancet. 2006 Jan 14;367(9505):133-43. doi: 10.1016/S0140-6736(06)67962-2. PMID 16413877
- [Result] Hadler MC, Sigulem DM, Alves Mde F, Torres VM. Treatment and prevention of anemia with ferrous sulfate plus folic acid in children attending daycare centers in Goiania, Goias State, Brazil: a randomized controlled trial. Cad Saude Publica. 2008;24 Suppl 2:S259-71. doi: 10.1590/s0102-311x2008001400011. PMID 18670706
- See also: Publication of the article — http://www.scielo.br/pdf/csp/v24s2/11.pdf
- See also: Erratum of the title — http://www.scielo.br/pdf/csp/v24n11/30.pdf